CLINICAL TRIAL: NCT04476615
Title: Effects of Fasting-mimicking Diet on Central and Peripheral Components of Fatigue, Muscular Resistance
Acronym: FMD_Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Matteo Bertucco, Associate Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 140166
Record Dates: First submitted 2020-07-07; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Fatigue; Muscle, Heart; Fasting; Diet, Healthy; Fatigue, Mental
Keywords: fatigue; fasting-mimicking diet; healthy; young adults; exercise
MeSH Terms: conditions — Fatigue; Fasting; Mental Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FMD (Experimental): Fasting-Mimicking diet (ProLon®)
  Interventions: Dietary Supplement: Fasting-Mimicking Diet (ProLon®)
- Placebo (Placebo Comparator): Low-energy bars (L-Nutra®) supplementation
  Interventions: Dietary Supplement: Placebo bars

INTERVENTIONS:
Dietary Supplement: Fasting-Mimicking Diet (ProLon®) — Dietary restriction: Fasting-Mimicking Diet (ProLon®). 5-days cycles spaced at 1-month intervals for 3 months (3 cycles in total).
  Other Names: Dieta Mima Digiuno® (italian name)
  Arms: FMD
Dietary Supplement: Placebo bars — Dietary supplementation: Low-energy bars (L-Nutra®) to integrate the daily nutritional habits - one bar per day.
  5-days cycles spaced at 1-month intervals for 3 months (3 cycles in total).
  Arms: Placebo

SUMMARY:
The aim of the study is to test a Fasting Mimicking Diet (FMD) for its efficacy on improving muscular resistance and endurance. The investigators will perform a randomized clinical trial to test the efficacy of the FMD on improving muscular strength, muscular resistance and endurance in physically active young adults (18-40 years of age). The study will include two arms: Placebo (Placebo diet) and FMD (3 cycles of 5-day fasting-mimicking diet within two months). Study endpoints will include muscular strength evaluation of lower limbs, cardio-pulmonary responses, neuromuscular function and muscle architecture. Subjects will be evaluated 4 times within 3 months: at baseline (T1), after the 1st cycle of diet (T2), 7 to 15 days after the 3rd cycle of diet maintaining baseline intensity (T3) and with re-assessment of Peak Power Output (T4).

ELIGIBILITY:
Inclusion Criteria:

* Male sex;
* Age Range: 18-40 years old;
* Body Mass Index (BMI) range between 18.5 and 30;
* METs minutes per week - calculated by International physical activity questionnaire (IPAQ) - between 600 and 3000.

Exclusion Criteria:

* Female sex;
* History of muscle, joints and nerves injuries to the upper and/or lower limbs in the previous 12 months;
* Body Mass Index (BMI) below 18.5 and above 30;
* METs minutes per week - calculated by International physical activity questionnaire (IPAQ) - below 600 or above 3000.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Difference in time to exhaustion (TTE) | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Difference between time points in time duration [s] of the exercise at a given power output (85%) and cadence (60 RPM), before the given work rate could not be sustained.
Change in maximal voluntary contraction (MVC) | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Variation between time points in maximal force voluntarily produced by the knee extensor muscles pre- and immediately post exercise, considering for lever length [N*m].
Change in voluntary (muscle) activation (VA) | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Change between time points in the percentage of muscle activated by volition. [%] To quantify voluntary activation, the amplitude of the superimposed twitch is expressed as a fraction of the twitch evoked by the same stimulus in the relaxed muscle.
Change in resting twitch force (RT) | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Force elicited at rest by electrical stimulation of the femoral nerve, considering for lever length [N*m].
Change in oxygen consumption (VO2) | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Variations of mean oxygen consumption at rest and at each minute while exercising (performance test).
Change in peak (task-specific) oxygen consumption (VO2) | baseline (T1) and after 2 months (T4).
  Peak oxygen consumption during the incremental test (maximal value during a 30" time-window).
Change in femoral (artery) blood flow (FBF) | at rest and during the performance test. Differences between each time point will be assessed: baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Measurements of common femoral arterial blood velocity (Vmean) and vessel diameter will be performed using ultrasound Doppler, distal to the inguinal ligament and proximal to the bifurcation of the deep and superficial femoral arteries. (FBF = Vmean p (vessel diameter/2)^2 * 60)
Change in median frequency of the power spectrum density of EMG | during the performance test at each time point: baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  EMG signal from the vastus lateralis (VL) muscle was recorded throughout exercise to estimate the output of spinal motoneurons and the development of peripheral fatigue.

SECONDARY OUTCOMES:
Change in carbon dioxide (VCO2) production | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Variation of physiological production of CO2 at rest and while exercising measured by a breath-by-breath system [L/min].
Change in minute ventilation (VE) | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Difference in ventilatory response at rest and while exercising measured by a breath-by-breath system [L/min].
Change in heart rate (HR) | baseline (T1); day 5 (1°diet cycle - T1), after 2 months (T3 and T4)
  Difference in the cardiac response at rest and while exercising measured by a heart rate monitor system.
Change in Peak Power Output (Wpeak) | baseline (T1) and after 2 months (T4).
  Difference in maximal power [Watts] achieved (last completed 1-min step) during the incremental test sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertucco, PhD, Principal Investigator — Department of Neurosciences, Biomedicine and Movement Sciences - University of Verona
Locations (1):
- Department of Neurosciences, Biomedicine and Movement Sciences, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: Data will be available upon request to the corresponding author after publication of the original article.

REFERENCES:
- [Derived] Nardon M, Venturelli M, Ruzzante F, Longo VD, Bertucco M. Fasting-Mimicking-Diet does not reduce skeletal muscle function in healthy young adults: a randomized control trial. Eur J Appl Physiol. 2022 Mar;122(3):651-661. doi: 10.1007/s00421-021-04867-2. Epub 2022 Jan 16. PMID 35034194